CLINICAL TRIAL: NCT02150044
Title: A Clinical Study of the Acclarent Tympanostomy Tube Delivery System for the Treatment of Patients Requiring Tympanostomy Tube Insertion for Otitis Media
Brief Title: Acclarent Tympanostomy Tube Delivery System for the Treatment of Patients Requiring Tympanostomy Tube Insertion
Acronym: inVENT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Acclarent (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPR005008
Record Dates: First submitted 2014-05-27; First posted 2014-05-29 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Otitis Media
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tympanostomy tube (Experimental): Performance and safety of tympanostomy tube delivery system
  Interventions: Device: Acclarent Tympanostomy Tube Delivery System (TTDS).

INTERVENTIONS:
Device: Acclarent Tympanostomy Tube Delivery System (TTDS). — tympanostomy tube delivery system

SUMMARY:
This was a non-significant risk (NSR), prospective, multi-center, single arm clinical trial that aimed to evaluate safety and performance of the Acclarent Tympanostomy Tube Delivery System (TTDS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with either chronic otitis media with effusion (OME) or recurrent acute otitis media (AOM) and scheduled to undergo tympanostomy tube insertion

Exclusion Criteria:

* History of sensitivity or reaction to anesthesia chosen for the procedure
* Markedly atrophic, mono- or bimeric, severely retracted, atelectatic or perforated tympanic membrane
* Otitis externa
* Active acute otitis media
* Otitis media pathology requiring T-tubes
* Stenosed ear canal
* Anatomy that precludes sufficient visualization of and access to the tympanic membrane
* Anatomy that necessitates tympanostomy tube placement in the posterior half of the tympanic membrane

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-02; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kirkland, Washington, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each investigator was required to treat a minimum of two (2) subjects as lead-in procedures prior to enrolling subjects to the test cohort.
  Subjects enrolled to the lead-in cohorts were required to meet the same eligibility criteria and complete the same protocol-required procedures as the study cohort.
Period: Overall Study
Arm/Group | Tympanostomy Tube
Started | 29
Lead-In Subjects | 16
Study Cohort | 13
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population includes 16 lead-in subjects and 13 study cohort subjects
Arm/Group | Tympanostomy Tube
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.7 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 12
  More than one race | 0
  Unknown or Not Reported | 11
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Ear Outcome Success
Description: Ear Outcome Success is successful delivery of the tympanostomy tube (TT) across the tympanic membrane (TM) per ear. This endpoint was evaluated for the 13 study cohort subjects only (not the 16 lead-in subjects).
Time Frame: Day 0 (at procedure visit)
Measure: Number; unit: ears
Units Other Than Participants: ears
Arm/Group | Tympanostomy Tube
Number analyzed (Participants) | 13
Number analyzed (ears) | 25
ears | 21

2. Secondary Outcome: Procedure Success
Description: Procedure Success is the successful placement of any tympanostomy tube evaluated on a per subject basis. This endpoint was evaluated for the 13 study cohort subjects only (not the 16 lead-in subjects).
Time Frame: Day 0 (at procedure visit)
Measure: Number; unit: participants
Arm/Group | Tympanostomy Tube
Number analyzed (Participants) | 13
participants | 12

3. Secondary Outcome: Tube Retention
Description: Tube Retention is the presence of a TTDS-placed tympanostomy tube across the tympanic membrane (TM) at the Follow-Up visit evaluated by ear. This endpoint was evaluated for the 13 study cohort subjects only (not the 16 lead-in subjects).
Time Frame: 1 week
Measure: Number; unit: ears
Units Other Than Participants: ears
Arm/Group | Tympanostomy Tube
Number analyzed (Participants) | 13
Number analyzed (ears) | 21
ears | 21

ADVERSE EVENTS:
Time Frame: up to 1 week post procedure
Description: Adverse event report includes both study cohort and lead-in subjects
Arm/Group | Tympanostomy Tube
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 5/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tympanostomy Tube (N=29)
Occluded Tube (Ear and labyrinth disorders) | 2 (2)
Otalgia (Ear and labyrinth disorders) | 1 (1)
Tube Medialization (Ear and labyrinth disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days